CLINICAL TRIAL: NCT03975023
Title: Assessing Neurophysiological Markers of Brain Function: Investigating Event-Related Potentials and Eye-Tracking Measures in Hockey Players
Brief Title: Investigating Event-Related Potentials and Eye-Tracking Measures in Hockey Players
Status: Completed | Type: Observational
Sponsor: Frederick Carrick, PhD, FACCN (Other)
Collaborators: HealthTech Connex Inc. (Industry)
Responsible Party: Sponsor-Investigator, Frederick Carrick, PhD, FACCN, Prof Frederick R Carrick, Carrick Institute for Graduate Studies
Organization: Carrick Institute for Graduate Studies (Other)
Other Study IDs: Carrick-001
Record Dates: First submitted 2019-05-30; First posted 2019-06-05 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Healthy; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- hockey players: During each study visit, the participants will undergo the following procedures:
  * NeuroCatch Platform (NCP) assessment (only if participant meets NCP-specific criteria)
  * RightEye's eye-tracking battery
  * Highmark Interactive's EQ application
  * Cambridge Brain Science's neuropsychological tests
  Interventions: Device: NeuroCatch Platform (NCP)

INTERVENTIONS:
Device: NeuroCatch Platform (NCP) — The NCP plays a proprietary 6-minute auditory stimulus sequence of tones and words that elicit involuntary evoked responses in the brain. Tone stimuli elicit N100 and P300 responses, and spoken word pairs elicit N400 responses. The NCP proprietary software identifies the latency and amplitude (timing and size) of three selected ERPs. Latency and amplitude values are reported as empirical (measured) values.

SUMMARY:
Traumatic brain injury (TBI) is a health issue impacting athletes and no clinical treatment protocol, other than rest, is yet established. The efficacy of a treatment protocol relies on objective, physiological measures of brain function and ultimately a quantification of injury severity.

The present study aims to assess neurophysiological markers of auditory and visual measures of brain function using the NeuroCatch Platform and eye-tracking technology, respectively. The current gold standard of TBI evaluation, including cognitive and balance assessments, will also be captured.

ELIGIBILITY:
Inclusion Criteria:

* Any sex, 14-25 years old inclusively
* Attending the Creative Artists Agency LLC (CAA) hockey camp in July 2019
* Able to understand the informed consent/assent form, study procedures and willing to participate in study

NeuroCatch Platform-Specific Inclusion Criteria

* Able to remain seated and focused for 6 minutes
* Normal hearing capabilities

Exclusion Criteria:

• Unable to provide informed consent

NeuroCatch Platform-Specific Exclusion Criteria

* Clinically documented hearing issues (e.g. tinnitus, in-ear hearing problems or punctured ear drum)
* In-ear hearing aid or cochlear implant, hearing device
* Implanted pacemaker or defibrillator
* Metal or plastic implants in skull
* Exposed to an investigational drug or device 30 days prior to start in this study, or concurrent or planned use of investigational drug or device during hockey camp (July 7th - 13th 2019)
* Not proficient in English
* Previous exposure to the NeuroCatch™ Platform audio sequences in the last 6 months
* History of seizures
* Allergy to rubbing alcohol or EEG gel
* Unhealthy scalp (apparent open wounds and/or bruised or weakened skin)

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Up to 70 hockey players aged 14-25 years will be included in the study.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
ERP response size | 1 week
  amplitude in microvolts
ERP response timing | 1 week
  latency in milliseconds
Eye-tracking: target accuracy | 1 week
  distance in millimeters for each eye
Eye-tracking: speed | 1 week
  degrees per second

SECONDARY OUTCOMES:
Cognitive tests | 1 year
  Cognitive assessments will be captured using Cambridge Brain Sciences battery of neuropsychological tests (composite score) and Highmark Interactive's EQ app
Balance | 1 week
  Balance measured in seconds as captured by Highmark Interactive's EQ app

OTHER OUTCOMES:
Trends between outcome measures and demographics will be explored | 1 year
  Demographics include age, concussion history, and handedness

CONTACTS AND LOCATIONS:
Locations (1):
- The Carrick Institute, Cape Cañaveral, Florida, United States